CLINICAL TRIAL: NCT05489562
Title: Use of Intraoral Suction and Its Effects on Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Principal Investigator, Ravi Rasalingam, MD, Cardiologist, VA Boston Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1686683
Record Dates: First submitted 2022-06-10; First posted 2022-08-05 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Obstructive Sleep Apnea of Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Mouthguard (Other): Subjects wearing mouthguard to access tolerability and comfort of the device
  Interventions: Device: Intraoral Suction

INTERVENTIONS:
Device: Intraoral Suction — stabilization of the tongue using intraoral suctioning and its effects on sleep parameters in patients with obstructive sleep apnea (OSA).

SUMMARY:
To learn whether stabilization of the tongue using intraoral suction is tolerable and what effects this approach has on sleep parameters in obstructive sleep apnea.

DETAILED DESCRIPTION:
Patients who are newly diagnosed with moderate OSA or diagnosed with OSA in the past 5 years and who are not compliant with continuous positive airway pressure treatment will be identified from the Boston VA Healthcare Sleep Laboratory database and invited to participate in the study. Those patients interested in participating will be consented and then evaluated for adequate nasal patency and oral dentition to assess their eligibility for the study. This is a pilot study primarily assessing tolerability of using intraoral suction to stabilise the tongue at night as well as its effects on sleep parameters. Target enrollment is 40 patients. Those enrolled will have a digital intra-oral scan performed and a custom-fit mouthguard that can transmit low level intermittent suction fabricated. The participant will wear this mouthguard for up to five consecutive nights. They will complete a survey designed to assess tolerability following five nights of wearing the mouthguard. The participant will then have a two night in-hospital polysomnography performed one night with the mouthguard transmitting suction and a second night with no suction. The outcomes will be measured using the tolerability survey scores and the duration and quality of sleep as measured by polysomnography.

ELIGIBILITY:
Inclusion Criteria:

Age 18-80

Patients newly diagnosed with OSA (a diagnosis of OSA ≤6 months) who may or may not have started using their PAP yet

Patients diagnosed > 6 months but within the past 5 years who are not compliant with positive airway pressure treatment. Non compliance is defined as use of device for an average of <4 hours/night OR < 5 nights/week

An AHI, REI or RDI or any synonymous term for AHI in the moderate to severe range (15-60)

A body mass index (BMI) less than <=40 (BMI within 1 year of enrollment date)

Adequate dentition to support a dental retainer

Exclusion Criteria:

Evidence of central sleep apnea or concomitant sleep disorder other than OSA

Currently using MAD or other form of mouth prosthesis to treat OSA

Prior surgical treatment for OSA

History of anatomic nasal obstruction

Use of medications that may affect sleep (hypnotic medications for the treatment of insomnia)

Use of pacemaker or implantable cardioverter-defibrillator (ICD)

Immunocompromised (i.e., susceptible to infection)

Open soars/wounds in patient's mouth

Active alcohol abuse or IV drug use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients reporting adverse events related to use of intraoral suction to stabilize the tongue as assessed by a survey | Up to 16 weeks
  Tolerability and comfort will be assessed by a survey completed by each study subject. Number of patients reporting moderate or more severe pain related to use of intraoral suction to stabilize the tongue as assessed by a self-reported survey using a 5-point pain scale. The survey will be completed by each study subject after having worn the mouthguard for up to 5 consecutive nights in a row. Moderate to severe pain is classified as a score of 3 or higher.after their having worn the mouthguard for up to 5 consecutive nights in a row

SECONDARY OUTCOMES:
Effect on sleep duration | Up to 16 Weeks
  Change in sleep duration (minutes) with and without intraoral suction as measured by polysomnography
Effect on sleep quality | Up to 16 Weeks
  Change in percentage time in rapid eye movement (REM) with and without intraoral suction as measured by polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Rasalingam, MD, Principal Investigator — VA Boston Healthcare System
Locations (1):
- VA Boston Healthcare System, Jamaica Plain, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peppard PE, Young T, Barnet JH, Palta M, Hagen EW, Hla KM. Increased prevalence of sleep-disordered breathing in adults. Am J Epidemiol. 2013 May 1;177(9):1006-14. doi: 10.1093/aje/kws342. Epub 2013 Apr 14. PMID 23589584
- [Background] Young T, Finn L, Peppard PE, Szklo-Coxe M, Austin D, Nieto FJ, Stubbs R, Hla KM. Sleep disordered breathing and mortality: eighteen-year follow-up of the Wisconsin sleep cohort. Sleep. 2008 Aug;31(8):1071-8. PMID 18714778
- [Background] Lee CHK, Leow LC, Song PR, Li H, Ong TH. Acceptance and Adherence to Continuous Positive Airway Pressure Therapy in patients with Obstructive Sleep Apnea (OSA) in a Southeast Asian privately funded healthcare system. Sleep Sci. 2017 Apr-Jun;10(2):57-63. doi: 10.5935/1984-0063.20170010. PMID 28966740
- [Background] Rotenberg BW, Murariu D, Pang KP. Trends in CPAP adherence over twenty years of data collection: a flattened curve. J Otolaryngol Head Neck Surg. 2016 Aug 19;45(1):43. doi: 10.1186/s40463-016-0156-0. PMID 27542595
- [Background] Caldwell JA, Knapik JJ, Shing TL, Kardouni JR, Lieberman HR. The association of insomnia and sleep apnea with deployment and combat exposure in the entire population of US army soldiers from 1997 to 2011: a retrospective cohort investigation. Sleep. 2019 Aug 1;42(8):zsz112. doi: 10.1093/sleep/zsz112. PMID 31106808
- [Background] Colrain IM, Black J, Siegel LC, Bogan RK, Becker PM, Farid-Moayer M, Goldberg R, Lankford DA, Goldberg AN, Malhotra A. A multicenter evaluation of oral pressure therapy for the treatment of obstructive sleep apnea. Sleep Med. 2013 Sep;14(9):830-7. doi: 10.1016/j.sleep.2013.05.009. Epub 2013 Jul 17. PMID 23871259
- [Background] Sarmiento KF, Folmer RL, Stepnowsky CJ, Whooley MA, Boudreau EA, Kuna ST, Atwood CW, Smith CJ, Yarbrough WC. National Expansion of Sleep Telemedicine for Veterans: The TeleSleep Program. J Clin Sleep Med. 2019 Sep 15;15(9):1355-1364. doi: 10.5664/jcsm.7934. PMID 31538607
- [Background] Truong KK, De Jardin R, Massoudi N, Hashemzadeh M, Jafari B. Nonadherence to CPAP Associated With Increased 30-Day Hospital Readmissions. J Clin Sleep Med. 2018 Feb 15;14(2):183-189. doi: 10.5664/jcsm.6928. PMID 29351826
- [Background] Opportunities Missed to Contain Spending on Sleep Apnea Devices and Improve Veterans' Outcomes. Department of Veterans Affairs - Office of Inspector General; January 14, 2020 2020
- [Background] Leng Y, McEvoy CT, Allen IE, Yaffe K. Association of Sleep-Disordered Breathing With Cognitive Function and Risk of Cognitive Impairment: A Systematic Review and Meta-analysis. JAMA Neurol. 2017 Oct 1;74(10):1237-1245. doi: 10.1001/jamaneurol.2017.2180. PMID 28846764